CLINICAL TRIAL: NCT04114565
Title: The Santiago Immigrant Wellbeing Study (STRING): Prevalence of Mood Disorders Among Immigrants in Santiago, Chile
Brief Title: Prevalence of Major Depression Among Immigrants in Santiago, Chile
Acronym: STRING
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Principal Investigator, Antonia Errazuriz, Assistant Adjunct Professor, Pontificia Universidad Catolica de Chile
Other Study IDs: 17051004; 96875479 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Major Depressive Disorder
Keywords: prevalence; mood disorders; affective disorders; major depressive disorder; service use; migration health; global mental health
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The general aim of this study is to explore the prevalence of major depressive disorder and the use of mental health services in the immigrant populations in the Metropolitan Region of Santiago, Chile.

The hypotheses are:

1. A healthy immigrant effect will be observed in the studied population by which their prevalence of major depressive disorder will be lower than the prevalence in the general Chilean population.
2. A significant association will be observed between the loss of socio-economic position after migration and a greater probability of major depressive disorder.
3. A significant association will be observed between the report of victimization experience(s) in the previous year and a greater probability of major depressive disorder.
4. A significant association will be observed between financial difficulties and a greater probability of major depressive disorder.

The sampling framework of the Chilean National Institute of Statistics (INE) from the 2016 Census will be used for the purpose of this research. The sampling units are as follows:

1. Primary sampling units (PSUs): conglomerates or groups of adjoining houses, organized in spatial blocks (200 households on average)
2. Secondary sampling units (SSUs): individual households within each of the conglomerates selected in the first stage
3. Final sampling units: persons meeting the study's inclusion criteria Multi-stage random probability sampling involving a 3-stage sampling design will be used - first, the sampling of the primary sampling units (PSUs); second, the sampling of households within the selected PSUs and finally, the random sampling of a household member.

Participants (n=1,100) will then take part in a 45-minute interview. This interview will be a household survey using the modular version of the Composite International Diagnostic Interview (WHO-CIDI) looking at exploring a broad spectrum of factors traditionally associated with increased risk of affective disorders:

1. Sociodemographics
2. Finance
3. Variation in socioeconomic position
4. Experience of victimization
5. Discrimination
6. Experience of childhood adversity

ELIGIBILITY:
Inclusion Criteria:

* Country of birth other than Chile
* Time since arrival to Chile: 3 months

Exclusion Criteria:

* Unable to understand Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults residing in private households in the Metropolitan Region of Santiago, Chile who were born outside of Chile and have lived in the country for at least 3 months
Sampling Method: Probability Sample
Enrollment: 1092 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Major Depressive Disorder | baseline
  Assessed using the World Health Organisation Composite International Diagnostic Interview (WHO-CIDI)
Any affective/mood disorder | baseline
  Assessed using the WHO-CIDI
Suicidal ideation, plans and attempts | baseline
  Assessed using the WHO-CIDI
Depressive symptoms | baseline
  Assessed using the nine-item Patient Health Questionnaire (PHQ-9).
  The PHQ-9 score can range from 0 to 27, with the following severity scores: 0-4 None; 5-9 Mild; 10-14 Moderate; 15-19 Moderate to Severe; 20-27 Severe.
Anxiety symptoms | baseline
  Assessed using the Generalized Anxiety Disorder 7-item scale (GAD-7).
  The GAD-7 score can range from 0 to 21, with the following severity scores: 0-4 None; 5-9 Mild; 10-14 Moderate; 15-21 Severe.

SECONDARY OUTCOMES:
Mental wellbeing | baseline
  Assessed using the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS).
  The 14 Items are scored on a range from 1 to 5, providing a total score between 14 and 70 with higher values indicating higher mental well-being.
Mental health service use | baseline
  Assessed using items of the Services Module of the WHO-CIDI
Hazardous/harmful drinking | baseline
  Assessed using the Alcohol Use Disorders Identification Test (AUDIT)

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Errazuriz, PhD, Principal Investigator — Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: Yes
IPD (database, dictionary) will be made available to researchers upon request.
Supporting Information: Study Protocol
Time Frame: 3 years after data collection ends
Access Criteria: Researchers with interest in mental health, particularly migration mental health

REFERENCES:
- See also: ISRCTN registry — https://doi.org/10.1186/ISRCTN96875479